CLINICAL TRIAL: NCT06668883
Title: Novel Exhaled Breath Aerosol Collection Devices in Patients With Lower Respiratory Tract Infection - a Performance and Acceptability Study (Acronym: AeroCAP)
Brief Title: Novel Exhaled Breath Aerosol Collection Devices in Patients With Lower Respiratory Tract Infection - a Performance and Acceptability Study
Acronym: AeroCAP
Status: Completed | Type: Observational
Sponsor: Avelo AG (Industry)
Collaborators: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-01738
Record Dates: First submitted 2024-10-29; First posted 2024-11-01 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Pneumonia; Lower Respiratory Tract Infection (LRTI)
Keywords: Respiratory Tract Infections; Pneumonia; Communicable Diseases; Infections; Breath
MeSH Terms: conditions — Pneumonia; Respiratory Tract Infections; Communicable Diseases; Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Sputum collection for molecular analysis — Sputum collection to be used with syndromic multiplex PCR testing
Device: Breath and cough collection for molecular analysis — Breath and cough collection with two proprietary devices to be used with syndromic multiplex PCR testing

SUMMARY:
This study will assess the performance of two novel breath collection devices and their subsequent detection of respiratory pathogens compared to sputum samples in patients with lower respiratory tract infections.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand the scope of the study and provide written informed consent
* Age >18 years
* Speaking German or English
* Health status (assessed by study personnel at local site) well enough to use the breath collection devices
* Willing to provide all three study samples (sputum and two breath samples) required for the study
* Clinical diagnosis of a lower respiratory tract infection (LRTI) defined as:

  (i) New infiltrate (chest X-ray, ultrasound, or CT scan), and (ii) at least one clinical symptom suggestive of LRTI (fever ≥38°C, chills, new or worsening cough, new or worsening sputum production, new or worsening dyspnea, tachypnoea, chest pain)

Exclusion Criteria:

* Patients for whom the collection of all three study specimens within 48 hours of initiating antibiotic treatment is not feasible
* Patients with known cystic fibrosis or bronchiectasis
* Critically ill patients at the discretion of the investigator
* Patients on oxygen supplementation with a face mask, high-flow-oxygen, non-invasive or mechanical ventilation; oxygen supplementation via nasal cannula will be permitted.
* Patients with proven acute pulmonary embolism
* Patients with best supportive care
* Patients with severe hypoxemia (SpO2 <88%) despite oxygen supplementation
* Hospitalization within the last 14 days prior to admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults aged 18 and older admitted to the hospital with a clinical diagnosis of lower respiratory tract infection.
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2024-11-13 (Actual); Primary Completion 2025-05-21 (Actual); Study Completion 2025-05-21 (Actual)

PRIMARY OUTCOMES:
Pathogen Concordance | 6 months
  Overall percent agreement, negative percent agreement, and positive percent agreement between syndromic respiratory multiplex PCR results from breath samples and sputum samples.

SECONDARY OUTCOMES:
Usability | 2 days after sample collection
  Assess the usability of the breath collection devices and sampling procedures by gathering user feedback from patients using a multiple choice questionnaire. Ease-of-use questions will be assessed using a 5-point difficulty rating system. Additionally, the investigators will assess the proportion of participants able to complete the breath collections without any deviations.
Expanded user feedback | 2 days after sample collection
  A subset of patients and clinicians will be observed during the breath collection process. The investigators will gather the proportion of participants making errors during breath collections and documenting any common difficulties.
  User feedback data from a subset of patients and clinicians will be gathered via semi-structured interviews. Data will be assessed qualitatively for reported acceptability and user preferences.
Rates of indeterminate breath results | 6 months
  Proportion of breath samples with invalid and/or indeterminate syndromic respiratory multiplex PCR results

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Basel, Basel, Switzerland